CLINICAL TRIAL: NCT06748924
Title: Chronic Coronary Syndrome Snapshot Study
Acronym: C2S2
Status: Recruiting | Type: Observational
Sponsor: European Society of Cardiology (Network)
Responsible Party: Sponsor
Other Study IDs: 2024-A01053-44
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Chronic Coronary Syndrome
Keywords: Observational study; ESC Guidelines; Chronic Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Chronic Coronary Syndrome: The study will include patients who align with the criteria set by the 2019 ESC Guidelines on CCS and that have been receiving medical care in accordance with these guidelines across 5 broad CCS categories: i) patients with angina and/or dyspnoea, and suspected coronary artery disease; ii) patients with new onset of heart failure or reduced left ventricular function; iii) patients with a long-standing diagnosis of CCS (i.e., those with stabilized symptoms <1 year after an acute coronary syndrome or with recent revascularization, and those >1 year after initial diagnosis or revascularization); iv) patients with angina without obstructive disease in the epicardial coronary arteries (i.e., microvascular angina, vasospastic angina); v) asymptomatic subjects referred to screening for coronary artery disease.

SUMMARY:
The goal of this observational study is to evaluate the current adherence to the 2019 European Society of Cardiology (ESC) Guidelines on Chronic Coronary Syndrome among healthcare professionals and identify potential barriers and facilitators to guideline implementation in patients with Chronic Coronary Syndrome (CCS). The main questions it aims to answer are:

AIM 1 - Evaluate Adherence to the 2019 ESC Guidelines on CCS Among Healthcare Professionals: To comprehensively assess the extent to which healthcare professionals adhere to the 2019 ESC Guidelines on CCS. • SUB AIM 1.1 - Assess Variations in Adherence Across Healthcare Settings: Identifying variations in adherence patterns across different healthcare settings (e.g., primary care clinics, specialty hospitals, and other healthcare facilities) to shed light on the impact of resource availability on guideline implementation.

* SUB AIM 1.2 - Analyse Regional Variations: Identifying variations in adherence patterns across different countries or regions, to provide insights into the influence of healthcare systems, cultural factors, and regional disparities on guideline adherence.
* SUB AIM 1.3 - Examine Disparities in Guideline Adherence: Identifying variations in adherence patterns among different demographic groups of healthcare professionals, including gender, age, years of experience, and specialty, to shed light on potential inequities in guideline implementation and help tailor interventions accordingly.

AIM 2 - Identify Potential Barriers and Facilitators to Guideline Implementation:

Through data analysis, we aim to identify potential barriers that hinder guideline implementation and facilitators that promote adherence and offer actionable insights for improvement. These barriers and facilitators may encompass a wide range of factors, including knowledge gaps, resource limitations, organizational constraints, and patient-related variables.

• SUB AIM 2.1 - Equitable access to cardiovascular care: Identifying variations in adherence patterns across sex and ethnicity categories, with a special focus on minorities.

Participants will not have more interventions than their usual care.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) refers to the presence of atherosclerotic plaques in the coronary arteries, which can be non-obstructive or obstructive. It represents a major cause of morbidity, mortality, hospitalization and health expenditure in Europe.

The European Society of Cardiology (ESC) plays a pivotal role in advancing the field of cardiology by regularly updating and disseminating clinical practice guidelines. In 2019, the ESC released the latest iteration of its guidelines for the diagnosis and management of Chronic Coronary Sydrome (CCS).

The Chronic Coronary Syndrome Snapshot (C2S2) study aims to evaluate the current adherence to the 2019 ESC Guidelines on CCS among healthcare professionals and identify potential barriers and facilitators to guideline implementation.

The results can inform targeted interventions and educational programs aimed at enhancing adherence to the 2019 ESC guidelines for CCS, ultimately improving patient outcomes and the quality of care for individuals with CCS.

C2S2 will enrol adult patients who sign a written informed consent form and with confirmed or suspected diagnosis of CCS amoung these 6 following CCS categories: i) patients with suspected CAD and stable anginal symptoms and/or dyspnoea; ii) patients with new onset of heart failure or left ventricular dysfunction and suspected CAD; iii) asymptomatic and symptomatic patients with stabilised symptoms within one year after an acute coronary syndrome, or patients with recent revascularisation; iv) asymptomatic and symptomatic patients beyond one year after initial diagnosis or revascularisation; v) patients with angina and suspected vasospastic or microvascular disease; vi) asymptomatic subjects in whom CAD is detected at screening To ensure the representativeness of all the potential healthcare settings, not only hospitals but also outpatient clinics, primary care practices, and healthcare providers in the community will be involved.

The study is designed with 2 visits: one at enrollment and one follow up visit at 3 months to assess the current practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with angina and/or dyspnoea, and suspected coronary artery disease.
* Patients with new onset of heart failure or reduced left ventricular function.
* Patients within 1 year after an acute coronary syndrome or recent revascularisation.
* Patients beyond 1 year after initial diagnosis or revascularisation.
* Patients with Angina with No Obstructive Coronary Artery disease (ANOCA)(e.g., microvascular angina, vasospastic angina).
* Asymptomatic subjects referred for screening for coronary artery disease.

Exclusion Criteria:

* Patients with a recent acute coronary syndrome (defined as those within 1 month of a diagnosis of unstable angina, non-ST-segment elevation myocardial infarction or ST-segment elevation myocardial infarction).
* Patients with conditions unrelated to CCS that significantly limit their ability to participate in the study or interfere with the assessment of guideline adherence.
* Patients participating in any clinical study where the protocol recommends deviations from guidelines recommendations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients who align with the criteria set by the 2019 ESC Guidelines on CCS and that have been receiving medical care in accordance with these guidelines across 5 broad CCS categories:
  i) patients with angina and/or dyspnoea, and suspected coronary artery disease; ii) patients with new onset of heart failure or reduced left ventricular function; iii) patients with a long-standing diagnosis of CCS (i.e., those with stabilized symptoms <1 year after an acute coronary syndrome or with recent revascularization, and those >1 year after initial diagnosis or revascularization); iv) patients with angina without obstructive disease in the epicardial coronary arteries (i.e., microvascular angina, vasospastic angina); v) asymptomatic subjects referred to screening for coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate Adherence to the 2019 ESC Guidelines | From enrollment to the follow up visit at 3 months
  Evaluate Adherence to the 2019 ESC Guidelines on CCS Among Healthcare Professionals: To comprehensively assess the extent to which healthcare professionals adhere to the 2019 ESC Guidelines on CCS

SECONDARY OUTCOMES:
Assess Variations in Adherence Across Healthcare Settings | From the enrolment and until the follow up visit at 3 months
  Identifying variations in adherence patterns across different healthcare settings (e.g., primary care clinics, specialty hospitals, and other healthcare facilities) to shed light on the impact of resource availability on guideline implementation
Analyse Regional Variations | From the enrolment and until the follow up visit at 3 months
  Identifying variations in adherence patterns across different countries or regions, to provide insights into the influence of healthcare systems, cultural factors, and regional disparities on guideline adherence.
Examine Disparities in Guideline Adherence | From the enrolment and until the follow up 3 months
  Identifying variations in adherence patterns among different demographic groups of healthcare professionals, including gender, age, years of experience, and specialty, to shed light on potential inequities in guideline implementation and help tailor interventions accordingly.
Identify Potential Barriers and Facilitators to Guideline Implementation | From the enrolment and until the follow up 3 months
  Through data analysis, we aim to identify potential barriers that hinder guideline implementation and facilitators that promote adherence and offer actionable insights for improvement. These barriers and facilitators may encompass a wide range of factors, including knowledge gaps, resource limitations, organizational constraints, and patient-related variables.
Equitable access to cardiovascular care | From the enrolment and until the end of follow up at 3 months
  Identifying variations in adherence patterns across sex and ethnicity categories, with a special focus on minorities

CONTACTS AND LOCATIONS:
Locations (1):
- Erebouni Medical Center, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: Undecided